CLINICAL TRIAL: NCT02203474
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Group, Dose-Ranging Study of 3 Doses of Tiotropium Hydrofluoralkane (HFA) Breath Actuated Inhaler (BAI), Placebo HFA BAI, and Open-Label SPIRIVA® HandiHaler® (18 mcg) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study of 3 Doses of Tiotropium Hydrofluoralkane (HFA) Breath Actuated Inhaler (BAI), in Patients With Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TBB-COPD-20009
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Tiotropium HFA BAI 5 mcg (Experimental): 1 inhalation from each of 3 inhalers containing either Tiotropium HFA BAI 5 mcg or placebo daily
  Interventions: Drug: Tiotropium HFA BAI 5 mcg
- Tiotropium HFA BAI 10 mcg (Experimental): 1 inhalation from each of 3 inhalers containing either Tiotropium HFA BAI 5 mcg or placebo daily
  Interventions: Drug: Tiotropium HFA BAI 5 mcg
- Tiotropium HFA BAI 15 mcg (Experimental): 1 inhalation from each of 3 inhalers containing either Tiotropium HFA BAI 5 mcg or placebo daily
  Interventions: Drug: Tiotropium HFA BAI 5 mcg
- SPIRIVA HandiHaler (Active Comparator): 2 inhalations from one 18 mcg capsule daily
  Interventions: Drug: Tiotropium 18 mcg Capsule
- Placebo (Placebo Comparator): 1 inhalation from each of 3 inhalers containing either Tiotropium HFA BAI 5 mcg or placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium HFA BAI 5 mcg
  Arms: Tiotropium HFA BAI 10 mcg; Tiotropium HFA BAI 15 mcg; Tiotropium HFA BAI 5 mcg
Drug: Tiotropium 18 mcg Capsule
  Other Names: SPIRIVA HandiHaler
  Arms: SPIRIVA HandiHaler
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the superiority of tiotropium hydrofluoroalkane (HFA) breath actuated inhaler (BAI) to placebo HFA BAI following repeated, once-daily dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 40 to 80 years of age, as of the screening visit (SV), who have signed an informed consent prior to initiation of any study related procedures.
2. Diagnosis of COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines.
3. A measured post-bronchodilator (albuterol 360 mcg) forced expiratory volume in 1 second (FEV1) ≥30% and <80% of predicted normal at the SV. Predicted normal will be determined using National Health and Nutrition Examination Survey (NHANES) III standard values for Caucasians, African Americans and Mexican-Americans with adjustments to predicted values made for Asian American patients.
4. A measured post-bronchodilator (albuterol 360 mcg) FEV1/forced vital capacity (FVC) <0.70 at the SV.
5. A minimum body weight of 40 kg. (Note: For patients participating in the pharmacokinetic [PK] sub study a minimum body weight of 50 kg is required.)
6. If female, is currently not pregnant, breast feeding, or attempting to become pregnant (for 4 weeks before the SV and throughout the duration of the study), and is of non-childbearing potential, defined as:

   * ≥1 year post-menopausal (6 months of spontaneous amenorrhea is permitted, provided there is a local record of serum follicle stimulating hormone >40 mIU/mL and this is source documented) or
   * Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, salpingectomy, or hysterectomy)

   Or is of childbearing potential, has a negative serum pregnancy test, and is willing to commit to using a consistent and acceptable method of birth control, as defined below, for the duration of the study:
   * Systemic contraception used for ≥1 month prior to screening, including birth control pills, transdermal patch, vaginal ring, implants, or injectables or
   * Double barrier methods (spermicide with any of the following: condoms, cervical cap, diaphragm, and vaginal contraceptive film) or
   * Intrauterine device (IUD) with a low failure rate defined as <1% per year (use of copper IUDs is not acceptable) Or is of childbearing potential and is not sexually active, has a negative serum pregnancy test, and, in the event the patient becomes sexually active, is willing to commit to using a consistent and acceptable method of birth control, as defined above, for the duration of the study. At the discretion of the investigator, total abstinence is acceptable in cases where the age, career (eg, priest), lifestyle, and/or sexual orientation of the patient ensures compliance.
7. Current or ex-smoker with ≥10 pack-year smoking history (number of cigarette packs smoked per day multiplied by the number of years smoked; eg, 2 packs/day for 3 years equals a 6 pack-year history).
8. Patient is free of any other medical conditions or concomitant treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study.
9. Able to perform technically acceptable and reproducible spirometry per American Thoracic Society/European Respiratory Society (ATS/ERS) 2005 guidelines and study guidelines, as defined in the protocol and study reference manual; this includes able to tolerate withdrawal of applicable medications during required spirometry assessments.
10. Able to perform acceptable peak expiratory flow measurements.
11. Able to maintain records (patient daily diary) during the study period as required by the protocol.
12. Able to demonstrate the proper inhalation techniques required for correct use of all delivery devices (BAI and dry powder inhaler [DPI]) required in the study.
13. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and being compliant with all study requirements.

Exclusion Criteria:

Chronic Obstructive Pulmonary Disease

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the patient's last study related visit (for eligible patients only, if applicable).
2. Current evidence of a clinically significant or uncontrolled disease including, but not limited to: cardiovascular (eg, uncontrolled hypertension, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (eg, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal (eg, poorly controlled peptic ulcer, gastroesophageal reflux disease), or pulmonary (other than COPD such as asthma, sarcoidosis, non cystic fibrosis bronchiectasis, cystic fibrosis, bronchopulmonary dysplasia or a diagnosis of alpha 1 antitrypsin deficiency). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the patient at risk through participation, or which could affect the endpoint analysis if the disease/condition worsened during the study.
3. History of and/or current diagnosis of asthma.
4. History of a life-threatening COPD exacerbation - defined for this protocol as a COPD episode that required intubation or was associated with respiratory arrest.
5. Thoracotomy with pulmonary resection.
6. Current congestive heart failure, history or current evidence of myocardial infarction (within 1 year of the SV), or current history of active ischemic heart disease (exertional or intermittent angina).
7. History or current evidence of clinically significant cardiac arrhythmia or abnormality, including a diagnosis on screening ECG. Findings that are always considered clinically significant and will exclude the patient from study participation include, but are not limited to, the following:

   * ventricular rate <45 beats per minute (bpm) or >100 bpm
   * PR interval >240 msec
   * evidence of 2nd- or 3rd-degree atrioventricular block (excluding MobitzI)
   * evidence of supraventricular or ventricular ectopy or arrhythmias
   * corrected QT interval (QTc) (Bazett's or Fridericia's method) >500 msec
   * nonspecific intraventricular conduction delay >120 msec
   * ST-T wave abnormalities (excluding nonspecific ST-T wave abnormalities) indicative of acute ischemia/infarction
   * right or left complete bundle branch block
   * artificial pacemaker
8. The patient has a medical condition that may potentially be aggravated by an anticholinergic drug such as tiotropium, eg:

   * The patient has a history or presence of glaucoma (particularly angle-closure glaucoma)
   * The patient has symptomatic prostatic hyperplasia.
   * The patient has a known history or any current evidence of renal impairment or urinary retention (eg, bladder outlet obstruction). This includes abnormal renal function test results at screening.
9. History of malignancy (excluding treated non-melanoma skin cancers) within the past 5 years, regardless of the clinical significance or current stability of the disease.
10. History of silent (or active) infections, including positive tests for human immunodeficiency virus (HIV) 1, HIV2, hepatitis B, hepatitis C, or tuberculosis.
11. Occurrence of any upper or lower respiratory infection, including but not limited to the common cold and flu, sinusitis, tonsillitis, pneumonia, bronchitis, or an ear infection (including otitis media and externa) which is not resolved by 4 weeks or more prior to the SV/informed consent.
12. Occurrence of a COPD exacerbation which is not resolved by 4 weeks or more prior to the SV/informed consent.

    • Note: An exacerbation of COPD is defined as any worsening of the patient's baseline COPD symptoms requiring any treatment beyond study medication, rescue albuterol or the patient's regular maintenance treatment. This includes requiring the use of systemic corticosteroids, antibiotics and/or emergency room visit or hospitalization.
13. Patients who require regular use of daytime oxygen therapy.
14. Patients who have started or stopped an exercise rehabilitation program within 4 weeks of the SV.
15. Known or suspected hypersensitivity or idiosyncratic reaction to tiotropium, or to any ingredients used in the study medication formulations.
16. Severe allergy to milk protein.
17. Significant adverse drug reactions, including allergy or hypersensitivity reactions, to atropine or any anticholinergic substance related pharmacologically to atropine (eg, ipratropium or oxitropium).
18. Use of any prohibited concomitant medications within the required (per protocol) washout periods prior to the SV.
19. Treatment with orally administered (excluding orally inhaled) β-adrenergic agonists (ie, oral albuterol).
20. Recent initiation of treatment or dose titration with β-adrenergic receptor antagonists (eg, non-selective β-receptor blocking agents such as β-blocking anti-hypertensive products) administered by any route. Permitted exceptions are: (1) Patients treated on a stable dose of non-selective β-receptor blocking agents for 3 months prior to SV or longer may be considered for enrollment if expected to maintain the same dose throughout the study and (2) Patients on a stable dose of cardioselective β1 adrenergic receptor antagonists (eg, atenolol, metaprolol, bisoprolol) for at least 1 week prior to the SV are permitted if expected to maintain the same dose throughout the study.
21. Treatment with drugs commonly recognized to prolong the QTc interval (eg, quinolones, amiodarone, disopyramide, quinidine, sotalol, chlorpromazine, haloperidol, ketoconazole, terfenadine, cisapride, and terodiline).
22. Treatment with strong cytochrome P450 (CYP) 2D6 or CYP3A4 inducers or inhibitors (eg, quinidine, ketoconazole and gestodene) within 30 days prior to the SV.
23. For patients using an inhaled corticosteroid, initiation or change in the dose of inhaled corticosteroids within the last 30 days prior to the SV, and/or the patient is not expected to maintain a stable dose of inhaled corticosteroids during the course of the study.
24. For patients using maintenance oral corticosteroids for COPD, the average daily dose should not be greater than10 mg of prednisone equivalent per day and the dose should have been stable over the 6 weeks prior to the SV. The patient's prior oral corticosteroid (OCS) dose should be maintained without change during the study. (Note that oral steroid bursts completed 6 weeks or more prior to screening are acceptable.)
25. Exposure to any investigational drug within 30 days or 6 half-lives (whichever is longer) prior to the SV.
26. Has a history of alcohol and/or substance abuse within the past 5 years. aa. Vulnerable patients (eg, persons kept in detention). bb. The patient is an employee of the study site or has an immediate family member or household member involved with the conduct of the study (including participation in the study).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-24 | Day 28

SECONDARY OUTCOMES:
FEV1 (AUC0-24) | Day 1
Trough FEV1 | Day 2
Percentage of patients with a COPD exacerbation | 28 Days
Percentage of Patients with Adverse Events | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.